CLINICAL TRIAL: NCT06272669
Title: Cumulative and Booster Effects of Multisession Prefrontal tDCS on Cognitive and Social Impairments in Adolescents With Autism Spectrum Disorder
Brief Title: Cumulative and Booster Effects of Multisession Prefrontal tDCS in ASD Adolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Yvonne Han, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: HSEARS20220216004
Record Dates: First submitted 2023-10-18; First posted 2024-02-22 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Transcranial Direct Current Stimulation; Autistic Spectrum Disorder; Electroencephalography
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: This study comprises 3 phases: Phase 1 will be a randomized controlled trial in which 90 participants will be randomly assigned to receive either active or sham-tDCS combined with computerized executive function training for 10 consecutive working days over 2 weeks period. The other 2 phases will be an open-label, crossover phase, in which for Phase 2, participants in the sham-tDCS group will receive 10-day active tDCS and assessments will be performed before and after the 10-tDCS session. Whereas bimonthly booster tDCS sessions will be provided to all tDCS responders for the first 3 months and monthly booster tDCS in the subsequent 3 months (Total 9 sessions in phase 3), and with assessments performed every month in Phase 3.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active-tDCS vs Sham-tDCS (Experimental): During the active- and sham-tDCS conditions, the participants will receive current with ramp up and ramp down mode for 10 seconds, eliciting a tingling sensation on the scalp that fades over seconds. Following that, the tasks will be initiated five minutes subsequent to the stimulation mode and terminated prior to its end for active-tDCS condition. Whereas, the sham condition with the same placement and intensity will only receive 30s initial stimulation and then discontinue. Throughout the active / sham-tDCS condition, participants are required to sit still and focus their attention on a "+" displayed on a computer monitor during the five-minute rest. After that, they will undergo active-tDCS (1mA, 20 min) to the left DLPFC or sham stimulation over 10 sessions in 2 weeks, while performing the executive function training tasks.
  Interventions: Device: Active-tDCS; Device: Sham-tDCS
- Crossover trial (Other): Participants in the sham-tDCS group will receive 10-day active tDCS and assessments will be performed before and after the 10-tDCS session.
  Interventions: Device: Active-tDCS
- Booster effect (Experimental): All tDCS responders (>10% reduction in SRS scores) will enrol on a 6 months follow-up phase in which they will be randomized to receive either bimonthly 20-minute booster tDCS sessions, or bimonthly 20-minute booster sham tDCS sessions for 3 months, followed by monthly 20-minute booster tDCS, monthly 20-minute booster sham tDCS, for another 3 months, with a maximum of 9 (sham) tDCS booster sessions.
  Interventions: Device: Active-tDCS; Device: Sham-tDCS

INTERVENTIONS:
Device: Active-tDCS — For active-tDCS condition, participants will receive stimulation on the dorsolateral prefrontal cortex with ramp up and ramp down mode for 10 seconds, eliciting a tingling sensation on the scalp that fades over seconds. Following that, a twenty-minute executive functional training task will be initiated five minutes subsequent to the stimulation mode, and the stimulation will be terminated when the training task ends.
Device: Sham-tDCS — For sham-tDCS condition, participants will receive initial stimulation with ramp up and ramp down mode for 30 seconds, eliciting a tingling sensation on the scalp then it will be discontinued. Participants will also receive the twenty-minute executive functional training task five minutes subsequent to the stimulation mode.
  Arms: Active-tDCS vs Sham-tDCS; Booster effect

SUMMARY:
Autism spectrum disorder (ASD) is a neurodevelopmental disorder characterized by disturbances in communication, poor social skills, and aberrant behavior. To date, ASD has no known cure, and the disorder remains a highly disabling condition. Recently, transcranial direct-current stimulation (tDCS), a non-invasive brain stimulation technique, has shown great promise as a potentially effective and cost-effective tool for reducing the core symptoms in patients with autism, such as anxiety, aggression, impulsivity, and inattention. Although the preliminary findings in patients with ASD are encouraging, it remains to be determined whether this experimental data can translate into benefits in real life. Further studies are needed to determine the factors that can lengthen the therapeutic effects or cognitive benefits of tDCS, and to determine possible risk factors associated with relapse in patients with ASD. Booster sessions of tDCS is an important component of treatment planning and prognosis and may promote better outcomes to control for resurgence of symptoms. This study has three aims. First, the investigators aim to evaluate the therapeutic effects of tDCS on improving cognitive function in patients with ASD. Second, the investigators aim to better understand the neural mechanisms underlying the neuro-enhancing effects of tDCS in patients with ASD. Third, the investigators aim to assess the effectiveness of booster treatment cycles of tDCS for enhancing cognitive and social functions in individuals with ASD.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are confirmed by a clinical psychologist based on the Diagnostic and Statistical Manual of Mental Disorders-5th Ed (DSM-V) criteria of Autism spectrum disorder and structured interview with their parents or primary caregivers on their developmental history using the Autism Diagnostic Interview-Revised (ADI-R).

Exclusion Criteria:

* Individuals without a confirmed diagnosis from the clinical psychologist, with a history of other neurological and psychiatric disorders and head trauma, or on psychiatric medication will be excluded from the study.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-06-02 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in social responsiveness - Social Responsiveness Scale-2nd edition (SRS-2) | Phase 1 (RCT): Week 0, week 2, week 4, and week 6 of the study (4 time points); Phase 2 (crossover): Week 0 and week 2 (2 time points); Phase 3 (follow-up): Week 6, 10, 14, 18, 22, 26 (6 time points)
  SRS-2 is a sensitive measure of social functioning in children that detects even subtle symptoms that are highly related to ASD. It uses a four-point scale and focuses on different aspects of socialization. The total score reflects the clinical effectiveness of tDCS, and higher scores indicate greater symptom severity. It has been shown that SRS-2 is sensitive to detect changes in social communication improvement related to improved cognitive functioning after treatment. SRS-2 assessments will be conducted 1 day before and 1 day after tDCS treatment.

SECONDARY OUTCOMES:
Clinical response in tDCS outcome | Phase 1 (RCT): Week 0, week 2, week 4, and week 6 of the study (4 time points); Phase 2 (crossover): Week 0 and week 2 (2 time points)
  Based on the tDCS outcome recorded 1 day after tDCS treatment, participants will be categorized into responders and non-responders based on the percentage of change in the total SRS score. Participants who show reductions of at least 10% in total SRS scores as compared to baseline scores will be considered responders. This percentage reduction benchmark was set with reference to the minimal clinically important difference (MCID) and calculated using the standard error measurement method from an ASD sample in a previous randomized controlled trial.
Change in neuropsychological measures - CANTAB® cognitive tests | Phase 1 (RCT): Week 0, week 2, week 4, and week 6 of the study (4 time points); Phase 2 (crossover): Week 0 and week 2 (2 time points); Phase 3 (follow-up): Week 6, 10, 14, 18, 22, 26 (6 time points)
  Cambridge Neuropsychological Test Automated Battery (CANTAB®) includes computerized tests that are correlated to neural networks and have demonstrated high sensitivity in detecting changes in neuropsychological performance. The tests in this battery-the Reaction Time (RTI), Spatial Working Memory (SWM), and Multitasking Tests (MTT)-are well validated and are highly sensitive to the core domains impaired in patients with ASD, including to response/reaction time, working memory, attention, inhibition, and cognitive flexibility.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hung Hom, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided